CLINICAL TRIAL: NCT03041649
Title: Mic-Key Versus Mini: A Prospective, Randomized Trial for Family Preference Comparing Low Profile Balloon Gastrostomy Buttons
Brief Title: Mic-Key Versus Mini One Family Preference Comparison
Acronym: MicKeyVMini
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16070489
Record Dates: First submitted 2017-01-09; First posted 2017-02-03 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Gastroesophageal Reflux; Feeding Disorder; Family Satisfaction
Keywords: Gastroesophageal Reflux; Feeding Disorder; Gastrostomy tube; Family Satisfaction; GT button; Enteral nutrition; Gastrostomy button
MeSH Terms: conditions — Gastroesophageal Reflux; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GT button change - Mic-Key (Active Comparator): Subjects randomized to the Mic-Key arm will have the Mic-Key button placed initially at surgery, and at the first gastrostomy change in the clinic at 2 months, will change to the Mini One button. At the routine 4-month visit, parents will be asked which button they prefer to keep.
  Interventions: Other: GT button change - Mini One
- GT button change - Mini One (Active Comparator): Subjects randomized to the Mini One arm will have the Mini One button placed initially at surgery, and at the first gastrostomy change in the clinic at 2 months, will change to the Mic-Key button. At the routine 4-month visit, parents will be asked which button they prefer to keep.
  Interventions: Other: GT button change - Mic-Key

INTERVENTIONS:
Other: GT button change - Mic-Key — After 2 months with each button, parents will be asked which button they prefer at the 4-month post-operational follow-up visit.
  Arms: GT button change - Mini One
Other: GT button change - Mini One — After 2 months with each button, parents will be asked which button they prefer at the 4-month post-operational follow-up visit.
  Arms: GT button change - Mic-Key

SUMMARY:
The objective of this study is to compare two low profile balloon gastrostomy button enteral feeding devices, both currently used as standard of medical care. The investigators aim to compare family preference and rate of complications between the two devices in a prospective cohort of children. This is the first step in comparing initial and long-term outcomes along with the need for seeking medical advice for gastrostomy site-related complications.

The secondary aim of this study is to follow this population long term (4 years) to document the prevalence of: granulation tissue, infection, skin breakdown, and how long the gastrostomy tube balloon remains functional (does not lose water).

DETAILED DESCRIPTION:
This is a single center prospective, randomized study with a crossover design, comparing two low profile balloon gastrostomy buttons (Figure 1), MIC-Key™ and MINI One™ that are routinely used at CMH. Each subject will be randomly assigned to one button type at the time of initial placement. After placement, standard practice is to perform the first gastrostomy change in the clinic at 2 months where the primary caregivers replace the button under supervision. Therefore, the initial device after randomization will remain in place for 2 months. At the first scheduled device change, the other type of button will replace the original gastrostomy button device. This will remain in place for another 2 months. At the routine visit at 4 months the parents will be asked to choose which button they prefer to keep. This will meet the primary outcome endpoint of the study. The investigators will continue to follow as many subjects as possible to 4 years in order to identify any potential differences in secondary end points.

A caregiver satisfaction survey is routinely used in the clinics. Parent responses to this survey will be also be used in the study analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 0-5 years of age requiring 0.8 cm or 1.0 cm gastrostomy feeding devices for enteral nutrition seen in the Surgery, GI or Special Care clinics
* Gastrostomy placement after IRB approval (enrollment will continue until 170 evaluable subjects have completed the 4 month visit. Expected attrition for the 4 year follow-up is 40%.
* English-speaking families

Exclusion Criteria:

* Children with dermatologic conditions influencing gastrostomy site healing and tract epithelialization
* Children with immunosuppression
* Children with active malignancy requiring treatment
* Inability to commit to 4 months follow up

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2016-11; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Parent preference | 4 months
  Parents will be asked which button they prefer to keep at the 4-month visit.

SECONDARY OUTCOMES:
Enteral Access Assessment Sheet | Up to 4 years after button placement
  Providers will complete a brief checklist of gastrostomy tube maintenance and site complications at the 2-month button change, 4-month visit, and all subsequent follow-up visits while the button while the G-tube remains in place.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelhadi RA, Dekonenko C, Dorman RM, Oyetunji TA, St Peter SD. A Prospective, Randomized Cross-over Trial of 2 Low-profile Gastrostomy Buttons to Determine Family Preference. J Pediatr Gastroenterol Nutr. 2020 Mar;70(3):386-388. doi: 10.1097/MPG.0000000000002585. PMID 31834114